CLINICAL TRIAL: NCT06322875
Title: A Prospective, Single-center, Randomized, Split-face Controlled, Single-blind Evaluation, Superiority Clinical Trial to Evaluate the Efficacy and Safety of RHC(III) for Injection Combined With SkinCeuticals RHC Serum.
Brief Title: A Clinical Study to Evaluate the Efficacy and Satisfaction of RHC Serum Combined With RHC(III) Injection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DeYi Aesthetic Medical Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKCCOL002
Record Dates: First submitted 2024-02-26; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Facial Wrinkles
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Side (Experimental): Each subject will randomly formulate the face on one side as the test side
  Interventions: Procedure: Recombinant type III humanized collagen solution for injection; Other: SkinCeuticals recombinant humanized collagen (RHC) serum; Other: Regular face cream smear
- Control Side (Placebo Comparator): Each subject will randomly formulate the face on one side as the control side
  Interventions: Procedure: Recombinant type III humanized collagen solution for injection; Other: Regular face cream smear

INTERVENTIONS:
Procedure: Recombinant type III humanized collagen solution for injection — Each subject will receive one injection of Recombinant type III humanized collagen solution for injection on the whole face
Other: SkinCeuticals recombinant humanized collagen (RHC) serum — Subjects received SkinCeuticals recombinant humanized collagen (RHC) serum application on the test side face
  Arms: Test Side
Other: Regular face cream smear — Subjects received Regular face cream smear application on the whole face

SUMMARY:
To evaluate the efficacy and safety of recombinant humanized collagen (type III) solution for injection combined with SkinCeuticals recombinant humanized collagen (RHC) serum Participants will be assessed by subjective questionnaire (FACE-Q Satisfaction with skin,Global Aesthetic Improvement Scale, et al) and some medical instruments (VISIA,Ultrascan UC22 et al)

DETAILED DESCRIPTION:
With the growth of photoaging and age, more people have the appearance of fine lines, skin laxity, roughness. Clinical evidences shown that RHC III injection can effectively improve fine line, skin plumpness and firmness to some extent; SkinCeutials RHC serum is capable of improving skin plumpness, firmness and elasticity, and improve rough skin condition.

A Prospective, single-center, randomized, split-face controlled, single-blind evaluation, superior efficacy clinical trial to evaluate the efficacy and safety of recombinant humanized collagen (type III) solution for injection combined with SkinCeuticals recombinant humanized collagen (RHC) serum, to explore the synergetic effects of injectable integrated skincare in Chinese population.

A total of 54 subjects will be enrolled in this study, and half of the face of each subject will be randomly assigned 1:1 to the test side and the control side.

The subjects will receive one injection of recombinant type III humanized collagen solution and will be followed up for 12 weeks after injection treatment.

Experimental group: SkinCeuticals RHC cream and Regular cream (twice daily) Control group: Regular cream (twice daily)

Participants will be assessed by subjective questionnaire (FACE-Q Satisfaction with skin,Global Aesthetic Improvement Scale, et al) and some medical instruments (VISIA,Ultrascan UC22 et al)

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30 and 55;
* According to the researchers' judgment, the subjects' facial skin is rough, dry and has obvious fine lines, and the Glogau photoaging rating is II to IV, which can be improved by treatment;
* Subjects voluntarily sign informed consent and agree to complete the follow-up prescribed by the trial.
* Note: All the above items are eligible for inclusion.

Exclusion Criteria:

* The subject has facial scars or skin diseases that may affect the judgment of the treatment effect, is in the stage of allergic attack, or has active infections (such as inflammatory acne, herpes simplex, etc.), and/or unhealed wounds, and is in the stage of progressive skin diseases such as vitiligo, psoriasis, etc.;
* had received or planned to have the following surgery or treatment prior to screening that affected the trial during the study period:

  1. Before screening or during the study period, it is planned to perform comprehensive surgical treatment for facial wrinkles, such as silicone, autologous fat transplantation, facial lift surgery, catch-line lifting, permanent dermal fillers (such as polymethyl methacrylate);
  2. Treatment with semi-permanent dermal fillers (e.g., L-lactic acid, hydroxyapatite, polycaprolactones, etc.) is planned for 18 months before screening or during the study period;
  3. Treatment with biodegradable dermal fillers (such as sodium hyaluronate gel or collagen) planned for 12 months prior to screening or during the study period;
  4. Screening 6 months before or during the study period is planned in the overall Department: Botulinum toxin, plastic therapy, energy equipment other than light conditioning therapy and intense pulse light (such as laser, radio frequency, ultrasound, etc.), skin grinding, chemical exfoliation of medium depth or greater depth or other exfoliative treatment (such as trichloroacetic acid, carbonic acid, 10% or more concentration of fruit acid or 2% or more concentration of salicylic acid, etc.);
  5. Light conditioning therapy, intense pulsed light, shallow exfoliation, or other exfoliative therapy (e.g., hydroxy acid at concentrations below 10% or salicylic acid at concentrations below 2%, etc.) are planned for 3 months prior to screening or during the study period;
* a history of multiple severe or hereditary allergies to any part of the body, who plan to undergo desensitization during the study period, or who are allergic to the ingredients of the drugs or devices used in the experimental treatment (hyaluronic acid, streptococcal protein, lidocaine or other amide anesthetics, etc.);
* the subject has a history of abnormal coagulation function, or has used or plans to use anticoagulation, antiplatelet, or thrombolytic therapy (e.g., warfarin, aspirin, etc.) within 14 days prior to screening;
* pregnancy or breastfeeding, planned pregnancy during the test, or positive pregnancy test results during the screening period;
* The subject has a history of serious diseases of major organs or active autoimmune diseases;
* Those with hypertrophic scars or cicatricial constitution;
* Participants who have participated in other clinical trials within 30 days prior to the screening period;
* The subject is judged by the investigator to have other systemic diseases that are not suitable for participation in the study;
* Subjects who are unable to communicate or do not follow instructions;
* Other conditions that the investigator considers inappropriate to participate in this experiment.

Note: All the above items are "no" to be selected

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
FACE-Q Satisfaction with skin | 4 weeks after injection
  FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after medical aesthetic treatment in the face.The PROM is used to assess the satisfaction skin care as well as its treatment on the patient's quality of life (QoL).
  The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better satisfaction

SECONDARY OUTCOMES:
Investigator Global Aesthetic Improvement Scale (I-GAIS) Rates | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 5-level scale ranging from "1" (very much improved) to "5" (very much worse) to determine the degree of improvement of the treated areas.
  the rates of I-GAIS was defined as the proportion of subjects with a GAIS score of 1-3.
Subject Global Aesthetic Improvement Scale (S-GAIS) Rates | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  Subject Global Aesthetic Improvement Scale (S-GAIS) is a 5-level scale ranging from "1" (very much improved) to "5" (very much worse) to determine the degree of improvement of the treated areas.
  the rates of S-GAIS was defined as the proportion of subjects with a GAIS score of 1-3.
Improvement rate assessed by Atlas | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  The investigator evaluated the improvement around the face using Atlas facial wrinkle atlas, a validated wrinkle scoring system, in which crow's feet were divided into 7 different grades, forehead wrinkles were divided into 9 grades, forehead fine lines were divided into 8 grades, and Yintang wrinkles were divided into 7 grades. A higher grade means more wrinkles.The improvement rate was defined as the proportion of subjects with at least 1 point reduction in the wrinkle rating in different regions.
Change in Cutometer® dual Analysis Score | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  The Cutometer® dual will be used to assess changes in skin outcomes. Analysis will be conducted by a board-certified dermatologist at baseline and follow up. Evaluated skin properties/parameters included skin moisture content, transepidermal water loss, skin elasticity, and skin tightness. Collection of these parameters will be performed using a probe dedicated to the Cutometer®dual. The results are then used to generate a comprehensive analysis report, which includes both the quantitative measurements and qualitative assessments, along with any corresponding scores or ratings assigned to different skin attributes.
Change in VISIA® Skin Analysis Score | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  VISIA® Skin Analysis system will be used to assess changes in skin outcomes. Analysis will be conducted by a board-certified dermatologist at Baseline and follow up. The VISIA® Skin Analysis system will be used to capture the images which will then be processed by the VISIA software.The software utilizes advanced algorithms to detect and measure specific skin attributes. The skin attributes/parameters evaluated will be spots, pores, wrinkles, texture (roughness and smoothness of the skin), purple patches of the dermal layer, brown patches of the dermal layer, red areas and porphyrins. These parameters are evaluated using the captured images and the specialized algorithms employed by the VISIA software. The results are then used to generate a comprehensive analysis report, which includes both the quantitative measurements and qualitative assessments, along with any corresponding scores or ratings assigned to different skin attributes.
FACE-Q Satisfaction with Outcome | Enrollment day, 2 weeks ±3 days after injection, 4 weeks ±5 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after medical aesthetic treatment in the face.The PROM is used to assess the perspective and impact of skin care as well as its treatment on the patient's quality of life (QoL).
  The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better outcome
FACE-Q Satisfaction with skin | Enrollment day, 2 weeks ±3 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after medical aesthetic treatment in the face.The PROM is used to assess the satisfaction skin care as well as its treatment on the patient's quality of life (QoL).
  The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better satisfaction
Change of the thickness and density of subjects' facial dermis | Enrollment day, 2 weeks ±3 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  Evaluation of the thickness and density of subjects' facial dermis. Subject will be submitted to the Ultrascan UC 22 equipment.

OTHER OUTCOMES:
Changes from baseline in skin uniformity and spot area ratio measurements collected by VISIA's face image acquisition instrument. | Enrollment day, 2 weeks ±3 days after injection, 8 weeks ±2 weeks after injection, and 12 weeks ±2 weeks after injection.
  VISIA® Skin Analysis system will be used to assess changes in skin outcomes. Analysis will be conducted by a board-certified dermatologist at Baseline and follow up. The VISIA® Skin Analysis system will be used to capture the images which will then be processed by the VISIA software.The software utilizes advanced algorithms to detect and measure specific skin attributes. The skin attributes/parameters evaluated will be skin uniformity and spot area ratio. These parameters are evaluated using the captured images and the specialized algorithms employed by the VISIA software. The results are then used to generate a comprehensive analysis report, which includes both the quantitative measurements and qualitative assessments, along with any corresponding scores or ratings assigned to different skin attributes.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolei Qin, Principal Investigator — DeYi Aesthetic Medical Clinic

IPD SHARING:
Plan to Share IPD: No
All data obtained during a clinical trial is owned jointly by the investigator and the clinical trial facility. Under the premise of mutual consultation, the clinical trial institution or the investigator decides to publish the research results.